CLINICAL TRIAL: NCT06937879
Title: Investigation of Factors Affecting Upper Extremity Function in Healthy Young Adults
Status: Completed | Type: Observational
Sponsor: KTO Karatay University (Other)
Responsible Party: Principal Investigator, Hasan Gerçek, Principle Investigator, KTO Karatay University
Other Study IDs: KaratayUH14
Record Dates: First submitted 2025-04-14; First posted 2025-04-22 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Function
MeSH Terms: interventions — Hand Strength

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Hand Grip Strength — The grip strength of the participants will be performed with a hydraulic hand dynamometer on a chair with back and arm support. The participant will be asked to squeeze the dynamometer with maximum force. The measurement will be performed 3 times and the average value will be recorded.

SUMMARY:
The aim of this study was to determine the effects of grip strength, motor imagery and two-point discrimination on upper extremity function in healthy young adults.

ELIGIBILITY:
Inclusion Criteria:

* Being a university student,
* Being between the ages of 18-35
* Not having any known upper extremity problems

Exclusion Criteria:

* Upper extremity surgery history
* Neurological problems
* Chronic diseases

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy young adults
Sampling Method: Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2025-04-21 (Actual); Primary Completion 2025-05-12 (Actual); Study Completion 2025-05-12 (Actual)

PRIMARY OUTCOMES:
Function | Baseline
  The Turkish version of the Shoulder, Arm and Hand Problems Questionnaire (DASH-T) will be used to assess the functional level of the upper extremity [10]. The DASH-T questionnaire consists of 30 questions. The first 20 questions ask about physical ability and the last 10 questions ask about pain and related functional and environmental limitations. As the score approaches zero, the functional level of the person is high; as the score moves away from zero, the functional level of the person is low.

SECONDARY OUTCOMES:
Grip strength | Baseline
  The grip strength of the participants will be performed with a hydraulic hand dynamometer on a chair with back and arm support. The participant will be asked to squeeze the dynamometer with maximum force. The measurement will be performed 3 times and the average value will be recorded.
Motor imagery | Baseline
  Motor imagery will be assessed through a left/right judgment task in which participants will be required to recognize whether hand images correspond to their left or right side using the Recognise™ application (Neuro Orthopaedic Institute, Adelaide, Australia). For this test, participants will be seated comfortably in front of a table, with both elbows flexed at 90◦ and both index fingers placed at the bottom of the screen of an electronic tablet. Multiple images of forearms (20 on each side) in multiple postures, angles and skin colors will be randomly displayed in the center of the screen of the device. Participants will be given standard instructions to decide as quickly and accurately as possible whether each image is of the right or left hand by clicking on the 'left' (left fingers) or 'right' (right fingers) buttons displayed at the bottom of the screen.
Two-point discrimination | Baseline
  Two-point discrimination will be assessed using a two-dot discriminator placed longitudinally and perpendicular to the index fingertip. The test score is the minimum distance at which the participant can discriminate between two dots in five consecutive trials. The assessment starts with a distance of 4 mm and is gradually reduced or increased depending on the participant's performance. A distance greater than 4 mm is considered impaired

CONTACTS AND LOCATIONS:
Locations (1):
- KTO Karatay University, Karatay, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No